CLINICAL TRIAL: NCT00343642
Title: Dietary Treatment of Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R21AT001628-01A2 (NIH); R21AT001628-01A2 (NIH)
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease; Inflammatory Bowel Disease
Keywords: Crohn's disease; Fructooligosaccharide; Inulin; Diet; Treatment; Bacterial flora; Oxidative stress
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Time; Diet

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Active Fructo-oligosaccharide (Experimental): Subjects received an active fructo-oligosaccharide supplement and a diet following the 2005 Dietary Guidelines for Americans.
  The fructo-oligosaccharide supplement was administered orally in a powder form two teaspoons daily.
  Interventions: Drug: Active fructo-oligosaccharide
- Placebo Fructo-oligosaccharide (Placebo Comparator): Subjects received a placebo fructo-oligosaccharide supplement and a diet following the 2005 Dietary Guidelines for Americans.
  Interventions: Drug: Placebo fructo-oligosaccharide
- Dietary Therapy (Active Comparator): Subjects received a placebo fructo-oligosaccharide supplement and a restrictive anti-inflammatory diet developed by the research team.
  Interventions: Dietary Supplement: Diet

INTERVENTIONS:
Drug: Active fructo-oligosaccharide — 2 teaspoons of active fructo-oligosaccharides daily and Time and attention administering usual dietary recommendations for a healthy diet based on 2005 Dietary Guidelines for Americans
  Other Names: Active fructooligosaccharide (FOS) and Placebo Diet; Time and Attention and Active Fructooligosaccharide
  Arms: Active Fructo-oligosaccharide
Drug: Placebo fructo-oligosaccharide — 2 teaspoons of placebo fructose powder ( to serve as the placebo equivalent of active treatment with fructo-oligosaccharides daily) and Time and attention administering usual dietary recommendations for a healthy diet based on 2005 Dietary Guidelines for Americans
  Other Names: Placebo Diet and Placebo Supplement; Tiem and Attention and Fructooligosaccharide Placebo
  Arms: Placebo Fructo-oligosaccharide
Dietary Supplement: Diet — A restrictive anti-inflammatory diet developed by the research team and 2 teaspoons of placebo fructose powder ( to serve as the placebo equivalent of active treatment with fructo-oligosaccharides daily)
  Other Names: Active Dietary Intervention and Placebo Supplement; Dietary Treatment and Fructooligosaccharide Placebo
  Arms: Dietary Therapy

SUMMARY:
Our objective is to determine whether a specific dietary intervention or a fructooligosaccharide (FOS) supplement has anti-oxidant or prebiotic effects and whether it is beneficial in the treatment of Crohn's Disease (CD.

DETAILED DESCRIPTION:
Several epidemiological studies and therapeutic observations in the complementary and alternative medicine (CAM) literature suggest that diet is key to development of CD and its treatment. The investigators took advantage of these CAM recommendations and designed dietary interventions. Our preliminary open label studies in IBD patients showed that our interventions are acceptable and well-tolerated and result in improvement, reducing symptoms and/or the degree of inflammation. The investigators are now seeking to validate this finding and determine the mechanisms underlying the effects of dietary manipulation-such as potential effects on colonic bacterial microflora. In another pilot study using 16s rDNA bacterial fingerprinting, the investigators demonstrated that the intestinal microflora of patients with CD differ significantly from healthy individuals. Whether the investigators can normalize/change the microflora of CD patients with dietary therapies, however, remains to be determined. Accordingly, the investigators designed a double blind placebo controlled study to test the hypotheses that: (1) dietary manipulation with either diet or a FOS supplement is an effective CAM therapy that prevents CD relapse (leads to maintenance of remission) and (2) such dietary manipulation can normalize the microflora of CD patients and decrease mucosal oxidative damage.

90 participants are expected to undergo the trial and have a 2:1 chance of receiving active therapy. The trial is seeking to enroll participants with inactive CD who have been medically induced into remission within 9 months of enrollment. Participants must be on their Crohn's medications at a stable dose for 3 months, which does not include steroids (e.g. Prednisone, Entocort) or antibiotics at the time of enrollment. Participants will be followed till relapse occurs or up to 52 weeks. Participants are asked to fill out a variety of questionnaires, keep a food and adverse event diary, and have a research, limited, unprepped flexible sigmoidoscopy for colonic tissue collection at the beginning and end of the study period.

Significance. This study could provide information to suggest diet or dietary supplement as a safe therapy for IBD and lay the groundwork for more definitive, randomized, controlled trials.

ELIGIBILITY:
Inclusion Criteria:

1. Documented ileocolonic or colonic CD based on classical history and classical endoscopic or surgical findings and histology compatible with CD;
2. Induction of remission with medical therapy within 9 months of the study;
3. Inactive CD for at least 2 weeks with CDAI score less than 150;
4. No change in IBD medication doses for 3 months;
5. No change in smoking habits a month prior to enrollment (because smoking may exacerbate CD) and acceptance of not-changing smoking habits during the term of the study).

Exclusion Criteria:

1. Patients with history of bowel obstruction and/or known strictures (as the high fiber content may precipitate obstruction);
2. Patients with extensive colonic or ileocolonic resection;
3. Patients with ileostomies or colostomies with diverted fecal stream;
4. Patients with isolated perianal/anorectal disease;
5. Patients with surgically induced remission;
6. Concomitant infection (e.g., C. difficile colitis);
7. Use of antibiotics within 4 weeks, or steroids, herbal remedies or diet therapies within 2 weeks of the onset of the trial or during the study;
8. Use of potential IBD exacerbators such as NSAIDs within 1 wk of the study;
9. Acute illness requiring immediate hospitalization for CD or other reasons;
10. Presence of symptomatic organic GI disease other than CD, hemorrhoids, hiatal hernia; GERD;
11. Pre-existent organ failure or severe comorbidities as these may change Gl flora:

    * Liver disease (cirrhosis or persistently abnormal AST or ALT that are 2X> normal);
    * Kidney disease (creatinine>2.0 mg/dL);
    * Uncontrolled psychiatric illness;
    * Clinically important lung disease or heart failure;
    * HIV disease;
    * Alcoholism;
    * Transplant recipients;
    * Patients receiving other immunosuppressant medications for comorbidities (e.g. Enbrel for rheumatoid arthritis);
12. Presence of short bowel syndrome or severe malnutrition with ideal body weight less than or equal to 90% or predicted;
13. Estimated survival <1 year and Karnofsky performance status <50%;
14. Desire to become pregnant during study or current pregnancy or nursing;
15. Desire to change smoking-status during the study;
16. Daily use of anticoagulation and antiplatelet medications;
17. Complicated IBD with anticipation of imminent surgical intervention during the term of the study;
18. Inability to have a regular follow-up and comply with study requirements.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2006-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ece A Mutlu, MD MBA, Principal Investigator — Rush University Medical Center; Ali Keshavarzian, MD, Study Director — Rush University Medical Center; Shahriar Sedghi, MD, Study Director — Gastroenterology Associates of Central Georgia
Locations (2):
- United States (2):
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Rush University Medical Center, Chicago, Illinois

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 54 subjects were randomized into a 12 month randomized, double blind, placebo controlled trial to test the efficacy of a specialized restrictive diet and a Fructo-oligosaccharide (FOS) supplement in maintenance of remission in patients with Crohn's disease (CD). Participants were recruited at Rush University, Chicago between Sept 2005-2012.
Groups:
- Time and Attention and Active Fructo-oligosaccharide: Subjects received an active prebiotic fructo-oligosaccharide supplement and a diet following the 2005 Dietary Guidelines for Americans
- Time and Attention and Fructo-oligosaccharide Placebo: Subjects received a placebo fructo-oligosaccharide supplement and a diet following the 2005 Dietary Guidelines for Americans.
- Dietary Therapy and Fructo-oligosaccharide Placebo: Subjects received a placebo fructo-oligosaccharide supplement and a restrictive anti-inflammatory diet developed by the research team.
Period: Overall Study
Arm/Group | Time and Attention and Active Fructo-oligosaccharide | Time and Attention and Fructo-oligosaccharide Placebo | Dietary Therapy and Fructo-oligosaccharide Placebo
Started | 19 | 19 | 16
Upto 3 Months Complete or Flare | 2 | 0 | 1
3-6 Months Complete or Flare | 4 | 2 | 2
Completed | 10 | 11 | 9
Not Completed | 9 | 8 | 7
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 4
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Flare up | 6 | 4 | 0

BASELINE CHARACTERISTICS:
Population: All participants were patients with Crohn's disease in remission.
Groups:
- Time and Attention + Active Fructooligosaccharide Supplement.: Time and attention + active fructooligosaccharide supplement.
  Time and attention + active fructooligosaccharide supplementation: 2 teaspoons of fructooligosaccharides daily
- Time and Attention + Fructooligosaccharide Placebo: Time and attention + fructooligosaccharide placebo
  Time and attention + fructo-oligosaccharide placebo: 2 teaspoons of placebo powder daily
- Dietary Therapy + Fructooligosaccharide Placebo: Dietary therapy + fructooligosaccharide placebo
  dietary therapy + fructo-oligosaccharide placebo: Medical nutrition therapy and 2 teaspoons of placebo powder
- Total: Total of all reporting groups
Arm/Group | Time and Attention + Active Fructooligosaccharide Supplement. | Time and Attention + Fructooligosaccharide Placebo | Dietary Therapy + Fructooligosaccharide Placebo | Total
Number analyzed (Participants) | 19 | 19 | 16 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 14 | 47
  >=65 years | 2 | 3 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.21 (12.43) | 48 (16.89) | 45.13 (14.17) | 45.46 (14.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 10 | 33
  Male | 9 | 6 | 6 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 5 | 0 | 5
  Not Hispanic or Latino | 19 | 14 | 16 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 4 | 2 | 4 | 10
  White | 15 | 16 | 12 | 43
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 19 | 16 | 54
Smoking [Number; unit: participants] — Participants were grouped as per their current smoking status.
  participants
    Smokers | 3 | 1 | 0 | 4
    Non-smokers | 16 | 18 | 16 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Flare Up of Crohn's Disease Through Month 12
Description: The efficacy of the dietary treatment was assessed by looking at the number of participants who flared.
Time Frame: Up to 12 months
Measure: Number; unit: participants
Arm/Group | Time and Attention + Active Fructooligosaccharide Supplement | Time and Attention + Fructooligosaccharide Placebo | Dietary Therapy + Fructooligosaccharide Placebo
Number analyzed (Participants) | 19 | 19 | 16
participants | 6 | 4 | 0

2. Primary Outcome: Quality of Life in Patients Taking Dietary Treatments
Description: Inflammatory Bowel Disease Questionnaire (IBDQ) overall scores at the exit visit of the study.It consists of 32 questons divided into four dimensions: bowel symptoms (10 items), systemic symptoms (5 items), emotional function (12 items) and social function (5 items). Every question has graded responses from 1 (worst situation) to 7 (best situation), and thus the total score is ranging from 32 to 224 with higher scores representing better quality of life.
Time Frame: At exit visit of study
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Time and Attention and Active Fructooligosaccharide Supplement: Subjects received an active prebiotic fructo-oligosaccharide supplement and a diet following the 2005 Dietary Guidelines for Americans.
- Dietary Therapy and Fructooligosaccharide Placebo: Subjects received a placebo fructo-oligosaccharide supplement and a restrictive anti-inflammatory diet developed by the research team.
Arm/Group | Time and Attention and Active Fructooligosaccharide Supplement | Time and Attention and Fructo-oligosaccharide Placebo | Dietary Therapy and Fructooligosaccharide Placebo
Number analyzed (Participants) | 19 | 19 | 16
units on a scale | 180.17 (24.78) | 197.42 (22.55) | 196 (18.52)

3. Primary Outcome: Safety of Dietary Treatments
Description: Data not collected
Time Frame: 90 days
Population: Data not Collected
Arm/Group | Time and Attention + Active Fructooligosaccharide Supplement | Time and Attention + Fructooligosaccharide Placebo | Dietary Therapy + Fructooligosaccharide Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Changes in Ileocolonic Flora
Description: Data not collected
Time Frame: 90 days
Population: Data not collected
Arm/Group | Time and Attention + Active Fructooligosaccharide Supplement | Time and Attention + Fructooligosaccharide Placebo | Dietary Therapy + Fructooligosaccharide Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Time and Attention + Active Fructooligosaccharide Supplement. | Time and Attention + Fructooligosaccharide Placebo | Dietary Therapy + Fructooligosaccharide Placebo
Serious Adverse Events (participants affected / at risk) | 2/19 | 1/19 | 0/16
Other Adverse Events (participants affected / at risk) | 19/19 | 19/19 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Time and Attention + Active Fructooligosaccharide Supplement. (N=19) | Time and Attention + Fructooligosaccharide Placebo (N=19) | Dietary Therapy + Fructooligosaccharide Placebo (N=16)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) — Participant had a syncopal episode (felt to be vasovagal) after a bowel movement at home. Participant had a history of vasovagal syncope before the trial. She fell and hit her head during the syncope and fully recovered. Was hospitalized overnight.
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Subject had cough fever and headache and was given Tamiflu for possible influenza. He developed nausea, vomiting possibly due to Tamiflu or infection and a fever of 103 degrees Fahrenheit. He was hospitalized for 3 days for IV fluids and antibiotics.
Crohn's flare up (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Subject presented with abdominal pain, diarrhea, nausea and vomiting felt to be either a Crohn's flare or a viral infection. She was hospitalized for 3 days. A colonoscopy revealed active Crohn's disease confirming a flare.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Time and Attention + Active Fructooligosaccharide Supplement. (N=19) | Time and Attention + Fructooligosaccharide Placebo (N=19) | Dietary Therapy + Fructooligosaccharide Placebo (N=16)
Cardio vascular and Pulmonary symptoms (Cardiac disorders) | 11 (13) | 9 (11) | 8 (14)
Endocrine signs and symptoms (Endocrine disorders) | 0 (0) | 3 (4) | 2 (2)
Allergy symptoms (Immune system disorders) | 3 (6) | 5 (6) | 4 (8)
Abnormal Heart exam (Cardiac disorders) | 0 (0) | 1 (1) | 3 (4)
Tooth issues (General disorders) | 0 (0) | 1 (1) | 1 (1)
Squamous cell skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
GenitoUrinary symptoms (Renal and urinary disorders) | 3 (8) | 3 (8) | 4 (4)
Fractures (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Fever (General disorders) | 6 (8) | 4 (4) | 3 (4)
Abnormal exam due to URI (Renal and urinary disorders) | 5 (6) | 7 (9) | 0 (0)
Joint pain/ MSK problems (Musculoskeletal and connective tissue disorders) | 12 (31) | 7 (29) | 9 (21)
Infection- GI (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Neurological symptoms (Nervous system disorders) | 12 (18) | 12 (17) | 6 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 5 (10) | 2 (2)
Infection- URI (Renal and urinary disorders) | 13 (31) | 9 (15) | 9 (20)
Nausea/Vomitting (General disorders) | 9 (16) | 4 (4) | 4 (4)
Eye symptoms (Eye disorders) | 0 (0) | 1 (2) | 3 (4)
Abnormal abdominal exam (Gastrointestinal disorders) | 8 (19) | 9 (20) | 4 (9)
Extraintestinal Symptoms of IBD other than arthritis /arthralgia (General disorders) | 1 (1) | 3 (5) | 4 (6)
Psychiatric symptoms (Psychiatric disorders) | 4 (4) | 7 (9) | 4 (6)
Infection-UTI (Renal and urinary disorders) | 0 (0) | 1 (3) | 1 (1)
GERD symptoms (Gastrointestinal disorders) | 5 (6) | 6 (8) | 0 (0)
Infection-Lip Herpes (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infection- HPV (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Diarrhea/Frequent BM (Gastrointestinal disorders) | 10 (14) | 6 (9) | 7 (8)
Perianal and Rectal pain/discomfort (Gastrointestinal disorders) | 0 (0) | 4 (7) | 2 (2)
Infection- Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection- Shingles (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Abdominal discomfort+pain (Gastrointestinal disorders) | 13 (57) | 13 (34) | 11 (37)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (6) | 2 (3) | 1 (1)
Infection- Genital (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Surgeries (Surgical and medical procedures) | 0 (0) | 3 (5) | 0 (0)
Skin lesions (Skin and subcutaneous tissue disorders) | 10 (14) | 7 (11) | 7 (10)
Decrease in Appetite (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 10 (13) | 4 (9) | 2 (3)
Gas/Flatus (Gastrointestinal disorders) | 7 (14) | 8 (11) | 5 (7)
Kidney Stone (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 3 (4) | 1 (2) | 0 (0)
Weight Decline (General disorders) | 0 (0) | 1 (2) | 1 (1)
Change in bowel habits (Gastrointestinal disorders) | 2 (3) | 2 (2) | 0 (0)
Urgency - Bowel (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1)
Tenesmus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hernia - abdominal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Weight Gain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Abnormal ear exam (Ear and labyrinth disorders) | 3 (4) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Portal Hypertension (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Pilot study, Slow recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No